CLINICAL TRIAL: NCT00561041
Title: Maintenance of Treatment Gains in Adolescents With Alcohol Related Disorders
Brief Title: Aftercare for Adolescents Treated for Alcohol Abuse and Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NIAAA_KAM_012187; NIH grant number RO1-AA012187
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol; alcohol use disorder; cognitive-behavioral therapy; brief phone aftercare intervention; individual aftercare therapy
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Brief phone aftercare intervention composed of 5 integrated cognitive-behavioral and motivational enhancement Therapies administered during a period of 3 months according to a similar schedule
  Interventions: Behavioral: Brief phone aftercare intervention
- 2 (Experimental): Individual aftercare therapy - composed of 5 integrated cognitive-behavioral and motivational enhancement Therapies administered during a period of 3 months according to a similar schedule
  Interventions: Behavioral: individual aftercare therapy
- 3 (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Brief phone aftercare intervention — Interventions is composed of 5 integrated cognitive-behavioral and motivational enhancement therapies administered during a period of 3 months according to a similar schedule
  Arms: 1
Behavioral: individual aftercare therapy — composed of 5 integrated cognitive-behavioral and motivational enhancement Therapies administered during a period of 3 months according to a similar schedule
  Arms: 2

SUMMARY:
The study examines the relative efficacy of two active aftercare interventions (i.e., face-to-face , brief phone) with no-active aftercare for adolescents who completed outpatient treatment for alcohol use disorders(AUD)

DETAILED DESCRIPTION:
In this study 177 adolescents meeting criteria for alcohol use disorders (AUD) received weekly cognitive-behavioral therapy group sessions. 144 completers were randomized into the 3 individual aftercare (AR) conditions noted above. Manualized active interventions were composed of 5 sessions of integrated motivational enhancement and cognitive behavioral therapies. Outcomes assessments were done at end of aftercare, 3-6-and 12 months post AC completion.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between the ages of 13-18 years
* Meeting criteria for DSM-IV alcohol use disorders
* Able to comprehend and read English at the 5th grade level
* Participant and family member are willing to provide a locator information.
* Not planning to move out of state during the next 12 months

Exclusion Criteria:

* Meet any substance dependence criteria other than nicotine or cannabis
* Meet life time diagnosis of schizophrenia
* Reported a suicidal ideation with a plan, suicidal attempt, or self-injurious behavior in the last 30 days
* Having a medical condition that may prevent them from consistently attending and constructively participating in treatment and aftercare

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 177 (Actual)
Dates: Start 2005-11; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Alcohol use (days of use and days of heavy drinking) | 3, 6, and 12 months post aftercare condition completion

SECONDARY OUTCOMES:
Drug use according to primary outcome timeframe | 3, 6, and 12 months post aftercare condition completion

CONTACTS AND LOCATIONS:
Overall Officials: Yifrah Kaminer, MD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States